CLINICAL TRIAL: NCT03077412
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled Study Evaluating the Efficacy and Safety of Filgotinib in the Treatment of Perianal Fistulizing Crohn's Disease
Brief Title: Study to Evaluate the Efficacy and Safety of Filgotinib in the Treatment of Perianal Fistulizing Crohn's Disease
Acronym: Divergence2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-419-4016; 2016-003153-15 (EudraCT Number)
Record Dates: First submitted 2017-03-08; First posted 2017-03-13 (Actual); Results first posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Fistulizing Crohn's Disease
MeSH Terms: interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Filgotinib 200 mg (Experimental): Filgotinib 200 mg + placebo to match filgotinib 100 mg for 24 weeks
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib
- Filgotinib 100 mg (Experimental): Filgotinib 100 mg + placebo to match filgotinib 200 mg for 24 weeks
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib
- Placebo (Experimental): Placebo to match filgotinib 200 mg + placebo to match filgotinib 100 mg for 24 weeks
  Interventions: Drug: Placebo to match filgotinib

INTERVENTIONS:
Drug: Filgotinib — Tablet(s) administered orally once daily
  Other Names: GS-6034; GLPG0634
  Arms: Filgotinib 100 mg; Filgotinib 200 mg
Drug: Placebo to match filgotinib — Tablet(s) administered orally once daily

SUMMARY:
The primary objective of this study is to evaluate the efficacy of filgotinib as compared to placebo in establishing combined fistula response at Week 24. Participants will have the option to enter a separate Long-Term Extension (LTE) study (GS-US-419-3896; NCT02914600) if they meet eligibility requirements.

ELIGIBILITY:
Key Inclusion Criteria:

* Males or non-pregnant, non-lactating females, ages 18 to 75 years, inclusive based on the date of screening visit
* Diagnosis of Crohn's disease (CD) with a minimum duration of CD of at least 3 months
* Has draining perianal fistulae as a complication of CD, confirmed by magnetic resonance imaging (MRI) at screening
* Previously demonstrated an inadequate clinical response, loss of response to, or intolerance of at least 1 of the following agents (depending on current country treatment recommendations/guidelines):

  * Antibiotics AND/OR
  * Immunomodulators AND/OR
  * Tumor necrosis factor α (TNFα) Antagonist
* Is willing and able to undergo MRI per protocol requirements
* Is willing and able to undergo flexible sigmoidoscopy per protocol requirements

Key Exclusion Criteria:

* Presence of current rectovaginal anovaginal or enterovesicular fistulae
* Presence of ulcerative colitis (UC), indeterminate colitis, ischemic colitis, fulminant colitis, or toxic mega-colon
* History of total proctocolectomy, total colectomy, presence of ileostomy or colostomy, or likely requirement for surgery during the study
* Use of any prohibited concomitant medications as described in the study protocol
* Active tuberculosis (TB) or history of latent TB that has not been treated

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (27):
- United States (13):
  - University of Miami Crohn's and Colitis Center, Miami, Florida
  - Center for Interventional Endoscopy - Florida Hospital, Orlando, Florida
  - University of South Florida South Tampa Campus, Tampa, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Louisville Clinical Trials Unit, Louisville, Kentucky
  - John Hopkins Gastroenterology and Hepatology Services at the Green Spring Station Clinic, Baltimore, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center - IBD Clinic, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - DHAT Research Institute, Garland, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - McGuire DVAMC, Richmond, Virginia
- Austria (2):
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Medical University of Vienna, Department of Internal Medicine III, Division Gastroenterology and Hepatology, Vienna
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- Canada (2):
  - Mount Sinai Hospital, Toronto
  - Toronto Digestive Disease Associates Inc., Toronto
- France (3):
  - CHU Grenoble Alpes - Hopital Michallon (main office), La Tronche
  - CHU de Rennes - Hôpital Pontchaillou (main office), Rennes
  - CHU Nancy - Hopital de Brabois, Vandœuvre-lès-Nancy
- Germany (2):
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Universitatsklinkum Jena, Jena
- Hungary (2):
  - Békés Megyei Központi Kórház Dr. Réthy Pál Tagkórháza, Békéscsaba, Bekes County
  - Bugát Pál Kórház, Gasztroenterológiai osztály, Gyöngyös, Heves County
- Istituto Clinico Humanitas, Rozzano, Italy
- Royal Devon and Exeter Hospital, Department of Gastroenterology, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reinisch W, Colombel JF, D'Haens GR, Rimola J, Masior T, McKevitt M, Ren X, Serone A, Schwartz DA, Gecse KB. Efficacy and Safety of Filgotinib for the Treatment of Perianal Fistulising Crohn's Disease [DIVERGENCE 2]: A Phase 2, Randomised, Placebo-controlled Trial. J Crohns Colitis. 2024 Jun 3;18(6):864-874. doi: 10.1093/ecco-jcc/jjae003. PMID 38366672

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe and the United States. The first participant was screened on 06 April 2017. The last study visit occurred on 17 February 2021.
Pre-assignment Details: 106 participants were screened. Participants who were non-responders, met disease worsening criteria or completed all procedures per protocol, were offered the option to continue into a separate Long Term Extension (LTE) study (GS-US-419-3896; NCT02914600), if deemed appropriate by the investigator.
Groups:
- Filgotinib 200 mg: Participants received filgotinib 200 milligrams (mg) and placebo to match (PTM) filgotinib 100 mg, once daily for 24 weeks.
- Filgotinib 100 mg: Participants received filgotinib 100 mg and PTM filgotinib 200 mg, once daily for 24 weeks.
- Placebo: Participants received PTM filgotinib 200 mg and PTM filgotinib 100 mg, once daily for 24 weeks.
Period: Overall Study
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Started | 17 | 25 | 15
Completed | 14 | 12 | 6
Not Completed | 3 | 13 | 9
Not completed — Non-Responder [Crohn's Disease Activity Index (CDAI) and Perianal CDAI non-response] at Week 10 | 1 | 5 | 3
Not completed — Protocol-Specified Disease Worsening | 1 | 3 | 3
Not completed — Adverse Event | 1 | 2 | 2
Not completed — Investigator's Discretion | 0 | 1 | 1
Not completed — Withdrew Consent | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Filgotinib 200 mg: Participants received filgotinib 200 mg and PTM filgotinib 100 mg, once daily for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo | Total
Number analyzed (Participants) | 17 | 25 | 15 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (11.2) | 41 (14.0) | 39 (11.8) | 40 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 4 | 23
  Male | 8 | 15 | 11 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of race information.
  Participants
    Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Race: Asian | 0 | 2 | 0 | 2
    Race: Black or African American | 1 | 2 | 1 | 4
    Race: Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0
    Race: White | 15 | 19 | 14 | 48
    Race: Other | 0 | 0 | 0 | 0
    Race: Not Permitted | 1 | 2 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of ethnicity information.
  Participants
    Ethnicity: Not Hispanic or Latino | 17 | 23 | 15 | 55
    Ethnicity: Hispanic or Latino | 0 | 1 | 0 | 1
    Ethnicity: Not Permitted | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 3 | 1 | 5
  Austria | 4 | 2 | 2 | 8
  Belgium | 1 | 1 | 1 | 3
  Hungary | 1 | 1 | 1 | 3
  United States | 4 | 15 | 8 | 27
  United Kingdom | 1 | 0 | 0 | 1
  Italy | 0 | 0 | 1 | 1
  France | 2 | 3 | 0 | 5
  Germany | 3 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Combined Fistula Response at Week 24
Description: Combined fistula response at Week 24 was defined as reduction of greater than or equal to (≥) 1 from baseline in the number of draining external perianal fistula openings that were present at baseline, and absence of fluid collections > 1 centimeter (cm) on magnetic resonance imaging (MRI) pelvis at Week 24, among participants with at least 1 draining external perianal fistula opening at baseline.
Time Frame: Week 24
Population: Participants in Full Analysis Set (all the randomized participants who received at least 1 dose of the study drug) with at least 1 draining external perianal fistula opening at baseline were analyzed.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 17 | 24 | 12
percentage of participants | 47.1 [26.0 to 68.9] | 29.2 [14.6 to 47.9] | 25.0 [7.2 to 52.7]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Test type: Superiority; Risk Difference in Percentages = 22.1, 90% CI 2-sided [-9.9 to 50.0] — The 90% exact confidence interval (CI) was calculated based on binomial distribution (Clopper-Pearson method)
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Test type: Superiority; Risk Difference in Percentages = 4.2, 90% CI 2-sided [-26.5 to 34.3] — The 90% exact CI was calculated based on binomial distribution (Clopper-Pearson method)

2. Secondary Outcome: Percentage of Participants Who Achieved Combined Fistula Remission at Week 24
Description: Combined fistula remission at Week 24 was defined as perianal fistula closure of all external openings that were draining at baseline, and absence of fluid collections > 1 cm on MRI of pelvis at Week 24, among participants with at least 1 draining external perianal fistula opening at baseline.
Time Frame: Week 24
Population: Participants in the Full Analysis Set with at least 1 draining external perianal fistula opening at baseline were analyzed.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 17 | 24 | 12
percentage of participants | 47.1 [26.0 to 68.9] | 25.0 [11.5 to 43.5] | 16.7 [3.0 to 43.8]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Test type: Superiority; Risk Difference in Percentages = 30.4, 90% CI 2-sided [-1.3 to 57.3] — The 90% exact CI was calculated based on binomial distribution (Clopper-Pearson method)
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Test type: Superiority; Risk Difference in Percentages = 8.3, 90% CI 2-sided [-22.5 to 38.1] — The 90% exact CI was calculated based on binomial distribution (Clopper-Pearson method)

3. Secondary Outcome: Time to Clinical Fistula Response up to Week 24
Description: Time to clinical fistula response was defined as the time interval in days from date of first dosing of study drug to the first observation (during scheduled or unscheduled clinical visits) when ≥ 1 of the draining external perianal fistula openings that were present at baseline achieves perianal fistula closure, among participants with at least 1 draining external perianal fistula opening at baseline. Participants not known to had a clinical fistula response were to have their clinical fistula response time censored at the last time that lack of clinical fistula response was documented.
Time Frame: Time from treatment start to first visit when ≥ 1 of the draining external perianal fistula openings that were present at baseline achieved perianal fistula closure up to Week 24
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 17 | 24 | 12
days | 15 [15 to 28] | 16 [15 to 71] | 35.5 [15 to 71]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.26, 90% CI 2-sided [0.64 to 2.49] — Hazard ratio was derived from Cox Proportional-Hazards model
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.90, 90% CI 2-sided [0.47 to 1.75] — Hazard ratio was derived from Cox Proportional-Hazards model

4. Secondary Outcome: Time to Clinical Fistula Remission up to Week 24
Description: Time to clinical fistula remission was defined as the time interval in days from date of first dosing of study drug to the first observation (during schedule or unscheduled clinical visits) of perianal fistula closure of all external openings that were draining at baseline, among participants with at least 1 draining external perianal fistula opening at baseline. Participants not known to had a clinical fistula remission were have their clinical fistula remission time censored at the last time that lack of clinical fistula remission was documented.
Time Frame: Time from treatment start to first visit when perianal fistula closure takes place of all external openings that were draining at baseline up to Week 24
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 17 | 24 | 12
days | 15 [15 to 70] | 29 [16 to 74] | 71 [26 to NA] — Not enough participants achieved clinical fistula remission to calculate upper 90% CI.
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.87, 90% CI 2-sided [0.87 to 4.01] — Hazard ratio was derived from Cox Proportional-Hazards model
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.37, 90% CI 2-sided [0.65 to 2.92] — Hazard ratio was derived from Cox Proportional-Hazards model

5. Secondary Outcome: Percentage of Participants Who Achieved Proctitis Remission at Week 24
Description: The simple endoscopic score for Crohn's disease (SES-CD) score evaluates 4 endoscopic variables (ulcer size, ulcerated surface, affected surface, and presence of narrowings). The total SES-CD is calculated as the sum of the 4 variables for the required bowel segment. Values are given to each variable and for every examined bowel segment. The SES-CD size of ulcer subscore ranges from 0 (none) to 3 (very large) and for ulcerated surface subscore ranges from 0 (none) to 3 (>30 % of affected area). Higher value of the subscore indicates disease worsening. Proctitis remission at Week 24 was defined as a proctitis SES-CD score (sum of ulcer size and ulcerated surface SES-CD endoscopy subscores for the rectum and anal canal) of 0 assessed by centrally read flexible sigmoidoscopy at Week 24, in participants that had moderately to severely active proctitis at baseline. Moderately to Severely Active Proctitis defined as proctitis SES-CD Score > 2.
Time Frame: Week 24
Population: Participants in the Full Analysis Set who had moderately to severely active proctitis at baseline were analyzed.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 10 | 13 | 7
percentage of participants | 10.0 [0.5 to 39.4] | 15.4 [2.8 to 41.0] | 28.6 [5.3 to 65.9]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Test type: Superiority; Risk Difference in Percentages = -18.6, 90% CI 2-sided [-55.6 to 21.3] — The 90% exact CI was calculated based on binomial distribution (Clopper-Pearson method)
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Test type: Superiority; Risk Difference in Percentages = -13.2, 90% CI 2-sided [-51.0 to 24.1] — The 90% exact CI was calculated based on binomial distribution (Clopper-Pearson method)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: First dose date up to 24 weeks plus 30 days; Adverse Events: First dose date up to 24 weeks plus 30 days
Description: All-Cause Mortality: All Randomized Set included all participants who were randomized in the study; Adverse Events: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Filgotinib 200 mg: Participants received filgotinib 200 mg and PTM filgotinib 100 mg, once daily for up to Week 26.
- Filgotinib 100 mg: Participants received filgotinib 100 mg and PTM filgotinib 200 mg, once daily for up to Week 29.3.
- Placebo: Participants received PTM filgotinib 200 mg and PTM filgotinib 100 mg, once daily for up to Week 27.9.
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/25 | 0/15
Serious Adverse Events (participants affected / at risk) | 5/17 | 2/25 | 1/15
Other Adverse Events (participants affected / at risk) | 13/17 | 14/25 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Filgotinib 200 mg (N=17) | Filgotinib 100 mg (N=25) | Placebo (N=15)
Crohn's disease (Gastrointestinal disorders) | 1 | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Suspected COVID-19 (Infections and infestations) | 1 | 0 | 0
Vulval abscess (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Filgotinib 200 mg (N=17) | Filgotinib 100 mg (N=25) | Placebo (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1
Photophobia (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 2 | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 2 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Crying (General disorders) | 0 | 0 | 1
Exercise tolerance decreased (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 0
Medical device pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Abscess (Infections and infestations) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 1 | 0
Abscess soft tissue (Infections and infestations) | 0 | 0 | 1
Anal abscess (Infections and infestations) | 3 | 0 | 1
Anal fungal infection (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 3 | 1 | 2
Nasopharyngitis (Infections and infestations) | 2 | 2 | 2
Oral herpes (Infections and infestations) | 2 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1
Mental impairment (Nervous system disorders) | 0 | 0 | 1
Taste disorder (Nervous system disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pharyngeal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/12/NCT03077412/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT03077412/SAP_001.pdf